CLINICAL TRIAL: NCT02561247
Title: Clinical Evaluation of the Prismaflex HF20 Set and Prismaflex® System 7.10 for Acute CRRT in Children
Brief Title: Prismaflex HF20 Set and Prismaflex® System 7.10/7.20 for Acute Continuous Renal Replacement Therapy (CRRT) in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gambro 1463
Record Dates: First submitted 2015-09-23; First posted 2015-09-28 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury in Pediatric Patients
Keywords: Acute Kidney Injury; Continuous Renal Replacement Therapy; Blood Urea Nitrogen (BUN); Prismaflex; Pediatric
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prismaflex HF20 CRRT (Experimental): Patients included in this arm will be treated for a minimum period of 20 of the first 24 hours and up to 72 hours with each Prismaflex® HF 20 Set with BUN, creatinine and bicarbonate being measured for statistical analysis at 12 hour intervals during CRRT treatment.
  Interventions: Device: Prismaflex HF20 CRRT Filter; Device: Prismaflex® System 7.10 and 7.20

INTERVENTIONS:
Device: Prismaflex HF20 CRRT Filter
Device: Prismaflex® System 7.10 and 7.20

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the Gambro Prismaflex® HF20 Set based on testing the hypothesis that it delivers sufficient renal replacement therapy to effectively treat acute kidney injury (AKI) in pediatric patients by reducing blood urea nitrogen (BUN).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a hospital admission body weight ≥8 and <20 kg (ie, ≥17.6 and <44.09 lbs).
2. Patients with AKI defined as either 1) AKI by the Kidney Disease Improving Global Outcomes (KDIGO) Acute Kidney Injury Guideline serum creatinine criteria, which is a >50% rise in serum creatinine over baseline or a 0.3 mg/dL SCr rise in 48 hours OR 2) as AKI by the Pediatric modified Risk, Injury, Failure, Loss, End-Stage Renal Disease (pRIFLE) criteria which is a 25% reduction in estimated creatinine clearance,16 OR 3) a serum creatinine >1.2 mg/dL. OR Patients with severe fluid overload, defined as a >10% fluid accumulation relative to the ICU admission.
3. Patients who have received RRT previously can be included in the study if >24 hours have elapsed since their previous RRT treatment.
4. Provide written informed consent from one or both parents, as required by the local IRB or legal guardians, unless one parent is deceased, unknown, incompetent or not reasonably available, or when only one parent has legal responsibility for the care and custody of the child per 21 CFR Part 50.55(e).

Exclusion Criteria:

1. Patients a) weighing 8.0-20.0 kg with a hemoglobin of <7.0 g/dL, b) weighing 8.0-12.0 kg with a hemoglobin of <8.0 g/dL (unless blood prime used), and c) weighing 12.1-20.0 kg with a hemoglobin of <7.5 g/dL (unless blood prime used).
2. Children who are wards of the state.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital Stanford, Stanford, California
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center of Dallas, Dallas, Texas
  - Seattle Children's Hospital - Divison of Nephrology, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Prismaflex HF20 CRRT: Patients included in this arm will be treated for a minimum period of 24 hours and up to 72 hours with each Prismaflex® HF 20 Set being measured for statistical analysis at 12 hour intervals during CRRT treatment.
Period: Overall Study
Arm/Group | Prismaflex HF20 CRRT
Started | 23
Completed | 17
Not Completed | 6
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Two filter changes required within the first 24 hours. | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was based on the intent-to-treat (ITT) principle and includes any patient who received CRRT on the Prismaflex HF20 Set for any period of time.
Arm/Group | Prismaflex HF20 CRRT
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: months] | 40.6 (21.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Black or African American | 3
  Asian | 3
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in BUN (mg/dL) at 24 Hours Following Initiation of CRRT
Description: Blood Urea Nitrogen (BUN)
Time Frame: 24 hours from CRRT initiation
Population: The full analysis set (FAS) was based on the intent-to-treat (ITT) principle and includes any patient who received CRRT on the Prismaflex HF20 Set for any period of time. Number of subjects (n=17) with evaluable data is shown, which is a subset of FAS (N=23).
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Prismaflex HF20 CRRT
Number analyzed (Participants) | 17
Percent Change | -58.118 (20.0848)
Statistical Analysis 1: Comparison: Prismaflex HF20 CRRT; P Value is from a one sample t-test compared against the null hypothesis value. No adjustments were made for multiple comparisons/multiplicity in this study, since there was only one primary endpoint, one arm, and one pre-specified primary null hypothesis; Test type: Other; p = 0.0008, t-test, 1 sided — P Value is from a one sample t-test compared against the null hypothesis value; Null Hypothesis Value = -38; Degrees of Freedom=16; t-value=-4.13

2. Secondary Outcome: Percent Change From Baseline in Creatinine (Umol/L) at 24 Hours Following Initiation of CRRT
Time Frame: 24 hours from CRRT initiation
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Prismaflex HF20 CRRT
Number analyzed (Participants) | 17
Percent Change | -45.687 (19.8848)

3. Secondary Outcome: Percent Change From Baseline in Bicarbonate (mmol/L) at 24 Hours Following Initiation of CRRT
Time Frame: 24 hours from CRRT initiation
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Prismaflex HF20 CRRT
Number analyzed (Participants) | 17
Percent Change | 38.287 (29.6885)

4. Secondary Outcome: HF20 Set Filter Survival Time
Description: Filters that were replaced any time CRRT was stopped for reasons other than the failure to mediate the two alarms specified were censored at their current duration of usage (filter clotted and TMP excessive). Only filters that were replaced due to the two alarms were considered events for this survival analysis. A total of 34 filters were used in the study and 22 filters were censored, leaving data from only 12 filters to complete the survival estimate. Due to the small amount of filter data available, only the 25th percentile survival estimate was used since the 50th and 75th percentiles were not reached. Filter life of filters were analyzed using a Kaplan Meier survival curve with quartile survival times after the start of CRRT.
Time Frame: Up to 72 Hours after Initiation
Population: FAS
Measure: Number (95% Confidence Interval); unit: hours
Units Other Than Participants: filters
Arm/Group | Prismaflex HF20 CRRT
Number analyzed (Participants) | 23
Number analyzed (filters) | 34
hours
  25th Percentile | 11.79 [5.07 to 68.09]
  50th Percentile | NA [18.65 to NA] — Due to the small amount of filter data available, only the 25th percentile survival estimate was used since the 50th and 75th percentiles were not reached.
  75th Percentile | NA [NA to NA] — Due to the small amount of filter data available, only the 25th percentile survival estimate was used since the 50th and 75th percentiles were not reached.

5. Other Pre Specified Outcome: Number of Participants Experiencing at Least One Prismaflex Alarms Related to Fluid Balance and Extracorpeal Life
Description: The end of the extracorporeal circuit life will be defined by the occurrence of one or both of the following Prismaflex ® System alarms, after which CRRT will be terminated and the extracorporeal circuit replaced:
  * Warning: Filter is Clotted, and/or
  * Caution: TMP (Trans Membrane Pressure) Excessive
  Alarms from Prismaflex ® System 7.10 related to fluid balance will be noted and recorded for the following alarms:
  * Caution: Flow Problem
  * Caution: Gain Limit Reached
  * Caution: Loss Limit Reached
Time Frame: Up to 72 hours from CRRT initiation
Population: FAS
Measure: Number; unit: participants
Arm/Group | Prismaflex HF20 CRRT
Number analyzed (Participants) | 23
participants
  Alarm: Warning Filter Clotted | 7
  Alarm: Caution TMP Excessive | 1
  Alarm: Caution Flow Problem | 13
  Alarm: Warning Loss Limit Reached | 0
  Alarm: Warning Gain Limit Reached | 0

ADVERSE EVENTS:
Time Frame: Up to 24 hours prior to CRRT (Screening) through HF20 CRRT End (72 hours), for a total of up to 96 hours
Arm/Group | Prismaflex HF20 CRRT
All-Cause Mortality (participants affected / at risk) | 2/23
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prismaflex HF20 CRRT (N=23)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Right Ventricular Failure (Cardiac disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Intraventricular Haemorrhage (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertensive Crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prismaflex HF20 CRRT (N=23)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
BRADYCARDIA (Cardiac disorders) | 3 (3)
HYPOTHERMIA (General disorders) | 4 (4)
HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 (2)
CITRATE TOXICITY (Injury, poisoning and procedural complications) | 2 (2)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 (6)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (3)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 2 (2)
AGITATION (Psychiatric disorders) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPERTENSION (Vascular disorders) | 4 (4)
HYPOTENSION (Vascular disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to significant enrollment challenges, the study was terminated early before achieving the planned number of patients enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter Healthcare Corporation reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT02561247/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT02561247/SAP_001.pdf